CLINICAL TRIAL: NCT03811873
Title: Assessment of Vertebral Fracture Risk Using VFA and Vertebral Strength Assessment With DXA-Finite Element Analysis in Liver Transplant Recipients in Pretransplant Period
Brief Title: Assessment of Vertebral Fracture Risk for First Time Liver Transplant Candidates
Acronym: VFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ejigayehu G. Abate, Assistant Professor of medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-004899
Record Dates: First submitted 2019-01-04; First posted 2019-01-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Metabolic Bone Disease; Transplant-Related Disorder; Secondary Osteoporosis
Keywords: transplant related disorders; liver transplant; transplant related bone disease
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Absorptiometry, Photon; Bone Density

STUDY DESIGN:
Intervention Model Description: Testing a single group of participants who are first time liver transplant candidates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vertebral fracture assessment (Other): Study participants undergoing evaluation for liver transplant and deemed to early for transplant will receive standard of care bone mineral density and vertebral fracture assessment..
  Interventions: Diagnostic Test: Dual x-ray absorptiometry; Other: Vertebral Fracture Assessment

INTERVENTIONS:
Diagnostic Test: Dual x-ray absorptiometry — DEXA is a means of measuring bone mineral density (BMD) using spectral imaging. Two X-ray beams, with different energy levels, are aimed at the bones. Soft tissue absorption is subtracted out, then the bone mineral density (BMD) can be determined from the absorption of each beam by bone.
  Other Names: DEXA; Bone mineral density
Other: Vertebral Fracture Assessment — Lumbar/thoracic spine x-ray and labs assessed for bone turnover markers.

SUMMARY:
The researchers are trying to compare the effectiveness of Vertebral Fracture Assessment (VFA) in addition to the current standard of care spine x-ray in evaluation pre-liver transplant patients.

ELIGIBILITY:
Inclusion criteria

* First time liver transplant candidates deemed too early for liver transplant
* 24 hour urine Creatinine clearance of > 40 mg/dl. However bone turnover markers (beta CTx and P1NP) will be measured only in those with creatinine clearance >60mg/dl

Exclusion criteria

* Patients with prior solid organ transplantation
* Liver/kidney combination will be excluded
* Patients with 24 hr. urine creatinine clearance < 40mL/minute
* Patients who have been on osteoporosis medications - Bisphosphonates [Fosamax (Alendronate), Actonel (Risedronate), Boniva (Ibandronate), or Reclast (Zoledronic acid)] Teriparatide (Forteo), Abaloparatide (Tymlos), Denosumab (Prolia), within the past 5 years
* Use of other systemic medications that can effect bone remodeling including sex hormone replacement therapy (estrogen or testosterone), calcitonin, androgen deprivation therapy, aromatase inhibitors, or SERMS in the past 6 months
* Underlying disease that significantly impacts bone metabolism such as primary hyperparathyroidism, hyperthyroidism, Paget's disease of bone, fibrous dysplasia, or malignancies with skeletal metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Incident of clinical fractures validated by spine x-ray or other imaging (vertebral fracture assessment -VFA) | 24 months
  Proportion of participants experiencing a clinical fracture validated by x-ray or other imaging (VFA) as compared to standard of care ( Spine X-ray)

SECONDARY OUTCOMES:
Changes in bone mineral density by dual x-ray absorptiometry | 24 months
  Bone mineral density changes seen in end stage liver disease in (grams/cm2) at baseline and 12 months
Percent changes from baseline to 12 months estimation of bone strength derived from finite element analysis | 24 months
  Bone strength measurements derived from finite element assessment changes from baseline to 12 months and correlation with clinical and radiographic risk of fracture
Changes in bone turnover markers in end stage liver disease | 24 months
  Bone turnover markers (Beta CTX, P1NP) percent changes from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ejigayehu G Abate, M.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials